CLINICAL TRIAL: NCT06170164
Title: Radiation Treatment of Lymph Node Recurrence From Prostate Cancer : is 11C-choline PET/CT Predictive of Survival Outcomes?
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: Colina-HTT-LN
Record Dates: First submitted 2023-11-28; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic accuracy — The aim of the study is to evaluate whether the pathological stage of the disease, Gleason score, age at diagnosis, serum PSA value and PET parameters (SUV, MTV) are predictive factors of choline PET examination.

SUMMARY:
The role of PET/CT with Choline in the restaging of prostatic disease is now universally recognized, and its use has become routine in numerous centers in Italy and abroad. The indication for the test is provided exclusively by an increase in PSA. It was interesting to understand whether these prognostic factors have an influence on the probability of detecting disease by PET with Choline to identify patients who have a greater probability of benefiting from the use of this method with the possibility of identifying the disease in earlier stages.

ELIGIBILITY:
Inclusion Criteria:

* patients operated with radical prostatectomy
* patients that present biochemical recurrence of the disease;

Exclusion Criteria:

* patients <18 years

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: The study is retrospective observational and the results of the choline PET diagnostic tests of 68 patients performed at our center from 2005 to 2013 were reviewed.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2015-11-25 (Actual); Study Completion 2015-11-25 (Actual)

PRIMARY OUTCOMES:
PET/CT with Choline in the restaging of prostatic disease. | 1 year
  retrospective analysis of 68 patients with biochemical recurrence of prostase disease that performed PET/CT with choline for the restaging of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: No